CLINICAL TRIAL: NCT07212634
Title: Efficacy and Mechanisms of Cerebellar Transcranial Direct Current Stimulation for Treating Dysphagia After Supratentorial Stroke
Brief Title: Cerebellar Transcranial Direct Current Stimulation for Dysphagia After Supratentorial Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Junmei Lai, MD, Attending Physician, Zhejiang Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024KY739
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Dysphagia After Stroke
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cerebellar tDCS Group (Experimental): This group will include 19 patients. The patients in this group will receive 20 minutes of tDCS over the bilateral cerebellar hemispheres.
  Interventions: Device: Transcranial Direct Current Stimulation
- Cortical (Suprahyoid Muscle) tDCS Group (Active Comparator): This group will include 19 patients. The patients in this group will receive 20 minutes of tDCS targeting the cortical representation areas of the suprahyoid muscles in both cerebral hemispheres.
  Interventions: Device: Transcranial Direct Current Stimulation
- Combined Cerebellar and Cortical (Suprahyoid Muscle) tDCS Group (Active Comparator): This group will include 19 patients. The patients in this group will receive 20 minutes of tDCS over the bilateral suprahyoid muscle cortical areas and 20 minutes over the bilateral cerebellar hemispheres.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS Group (Sham Comparator): This group will include 19 patients. The patients in this group received sham stimulation applied to the same area for the same duration.
  Interventions: Other: Sham tDCS

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Different experimental groups received tDCS stimulation at the following distinct sites: bilateral cerebellar hemispheres, bilateral cortical areas corresponding to the suprahyoid muscles, and combined bilateral cerebellar hemispheres alongside bilateral cortical areas corresponding to the suprahyoid muscles.
  Stimulation parameters: 2 mA constant current, 20 minutes per session Treatment regimen: 5 sessions per week for 2 consecutive weeks
  Arms: Cerebellar tDCS Group; Combined Cerebellar and Cortical (Suprahyoid Muscle) tDCS Group; Cortical (Suprahyoid Muscle) tDCS Group
Other: Sham tDCS — The patients in this group will receive sham stimulation applied to the same area for the same duration.
  Arms: Sham tDCS Group

SUMMARY:
It is estimated that 400,000 to 800,000 people worldwide develop neurogenic dysphagia annually. Stroke represents the most common etiology, with approximately 65% of acute stroke patients experiencing pharyngeal swallowing difficulties. Clinical manifestations of dysphagia vary widely in severity and may include residue, reflux, delayed swallowing initiation, aspiration, and cricopharyngeal muscle dysfunction. Due to its detrimental effects on nutrition, respiration, and psychosocial well-being, dysphagia significantly impairs patients' quality of life. Furthermore, the inability to swallow safely and efficiently can lead to serious complications such as aspiration pneumonia, malnutrition, and depression. The traditional swallowing rehabilitation treatment has limited effect in clinical practice, which makes it necessary to search for new effective swallowing methods.

Conventional swallowing rehabilitation often yields limited clinical benefits, highlighting the urgent need for more effective therapeutic strategies. Transcranial direct current stimulation (tDCS) is a non-invasive and safe neuromodulation technique that has shown promise in the field of neurorehabilitation. Its mechanisms extend beyond immediate cortical modulation and cerebral blood flow changes to include the regulation of synaptic plasticity, neurotransmitters such as glutamate and GABA, and excitability in remote subcortical regions. In recent years, tDCS has been increasingly applied to various neurological disorders, including post-stroke motor impairment, dysphagia, aphasia, depression, addiction, and spinal cord injury-related movement disorders. Currently, tDCS is being explored to elucidate its regulatory effects on cerebellar swallowing control, positioning it as a potential innovative treatment for neurogenic dysphagia.

DETAILED DESCRIPTION:
This multicentre randomized controlled trial will enroll 76 patients with dysphagia after stroke from Zhejiang Provincial People' s Hospital. All patients will be centrally randomized to either tDCS combined with traditional swallowing rehabilitation or traditional rehabilitation alone. The tDCS group will be further divided into three subgroups based on stimulation parameters. Observation indicators will be Standardized Swallowing Assessment (SSA), videofluroscopic swallowing study (VFSS) and neuroimaging examinations including fMRI, MRS And quantitative electroencephalography (QEEG).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with supratentorial stroke, confirmed by cranial MRI or CT as having cerebral infarction or hemorrhage;
2. Stable vital signs after conventional treatment, with disease duration between 1 and 6 months;
3. 30 ≤ age ≤75 years, male or female;
4. Presence of dysphagia, drinking-induced coughing, and a Kubota Water Drinking Test grade of 3-5;
5. Signed informed consent form.

Exclusion Criteria:

1. MRI-confirmed lesion involving the cerebellum;
2. Unstable vital signs;
3. Significant cognitive impairment (MMSE score ≤ 24);
4. Presence of swallowing apraxia;
5. Unwilling or unable to cooperate with treatment, or taking any medication that may affect swallowing function or nervous system activity.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized Swallowing Assessment (SSA) | at baseline (pre-treatment), at 2 weeks after intervention, at 3-month follow-up]
  Process: A clinician-administered scale performed in three sequential parts. Part 1 examines basic clinical signs (e.g., consciousness, lip closure, voluntary cough). Part 2 involves observing the patient swallowing 5ml of water three times. If no abnormalities are detected, Part 3 requires the patient to swallow 60ml of water, noting the time and signs of aspiration.
  Assessment: The total score (ranging from 18 to 46) is calculated. A higher score indicates more severe swallowing impairment.
Video fluroscopic swallowing study (VFSS) | at baseline (pre-treatment), at 2 weeks after intervention, at 3-month follow-up
  Process: Patients will swallow barium-coated boluses of varying consistencies (liquid, semi-solid) under real-time X-ray (videofluoroscopy). The procedure is recorded for frame-by-frame analysis.
  Assessment: The primary metric from VFSS will be the Penetration-Aspiration Scale (PAS ) score, which quantifies the depth and patient response to airway invasion. Additionally, the Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) scale or component scores for oral and pharyngeal phase efficiency and safety may be used. A lower PAS score indicates better airway protection.

SECONDARY OUTCOMES:
Change in Surface electromyography (sEMG) | at baseline (pre-treatment), at 2 weeks after intervention, at 3-month follow-up
  Process: Electrodes will be placed on the skin overlying the submental muscle group (suprahyoid muscles). Patients will perform swallowing tasks (e.g. saliva swallow, water swallow) while the electrical activity of these muscles is recorded.
  Assessment:
  1. Submental Electromyography (sEMG) Peak Amplitude (microvolts, µV): An indicator of the intensity of muscle contraction during swallowing, reflecting the degree of muscle effort.
  2. sEMG Burst Duration (milliseconds, ms): The time interval from the onset of muscle activation to its return to baseline levels, reflecting the coordination and efficiency of the swallowing act.
  3. sEMG Swallowing Waveform Morphology: The overall shape and pattern of the electrical activity signal during swallowing (e.g. a smooth, single-peak curve vs. a fragmented, multi-peak curve), used to assess the coordination of neuromuscular control. Changes in these parameters reflect improvements in the coordination and efficiency of the swallowing musculature.
Change in Functional magnetic resonance imaging (fMRI) | at baseline (pre-treatment), at 2 weeks after intervention, at 3-month follow-up
  Process: Using a 3.0T MRI scanner, high-resolution T1-weighted anatomical images and resting-state fMRI (rs-fMRI) data will be acquired. During rs-fMRI, patients will remain awake, relaxed, and with their eyes open, without performing any specific task.
  Assessment: Analysis will focus on changes in functional connectivity (FC) within the swallowing network, particularly between the cerebellum, primary sensorimotor cortex, and brainstem. Regional changes in the amplitude of low-frequency fluctuations (ALFF) or cerebral blood flow (CBF) will also be examined to identify alterations in local neural activity.
Change in Magnetic resonance spectroscopy (MRS) | at baseline (pre-treatment), at 2 weeks after intervention, at 3-month follow-up
  Process: A single-voxel MRS sequence will be performed. Voxels will be placed in key regions of interest (ROIs), including the bilateral swallowing motor cortex and the cerebellar hemispheres.
  Assessment: The concentrations of key neurometabolites-N-acetylaspartate (NAA, a marker of neuronal integrity), Choline (Cho, related to membrane turnover), Creatine (Cr, an energy reference), Gamma-Aminobutyric Acid (GABA, the primary inhibitory neurotransmitter), and Glutamate (Glu, the primary excitatory neurotransmitter)-will be quantified. Changes in ratios (e.g., NAA/Cr) or absolute concentrations will indicate neuroplastic and neurochemical changes.
Change in Quantitative electroencephalography (QEEG) | at baseline (pre-treatment), at 2 weeks after intervention, at 3-month follow-up
  Process: A 32-channel digital EEG system will record brain electrical activity for at least 10 minutes in a resting state (eyes closed). Data will be carefully inspected to remove artifacts.
  Assessment: The power spectral density of key frequency bands (Delta, Theta, Alpha, Beta) will be analyzed. Primary QEEG metrics will include the Brain Symmetry Index (BSI) to assess interhemispheric balance and the Delta + Theta/Alpha+Beta Ratio (DTABR), which serves as an indicator of overall brain arousal and cortical inefficiency. A decrease in DTABR suggests a shift towards a more alert and efficient brain state.

IPD SHARING:
Plan to Share IPD: No